CLINICAL TRIAL: NCT04238520
Title: Functionally-tailored Oral Care Intervention for Community-dwelling Older Adults With Dementia and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xi Chen (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor-Investigator, Xi Chen, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201803835; R21NR017347 (NIH)
Record Dates: First submitted 2020-01-10; First posted 2020-01-23 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Dementia; Cognitive Impairment
Keywords: Dementia; Caregiver; Family Relations; Oral Hygiene; Cognitive Impairment; Functional Level; Oral Health Education
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: control vs. intervention
Who Masked: Investigator
Masking Description: Single Blind- Study participants will be aware of the treatment assigned. The investigator and statistician will not know the group allocation. To check the success or failure of the blinding, the oral examiners and data collectors will be asked after each assessment whether they have been told or know for sure to which group each dyad has been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): PWD/CG dyads
  Interventions: Behavioral: Control Intervention
- Interventional (Experimental): PWD/CG dyads
  Interventions: Behavioral: Functionally Tailored Oral Care Intervention

INTERVENTIONS:
Behavioral: Functionally Tailored Oral Care Intervention — Participants receive a 4-week, hands-on, functionally-tailored intervention. The intervention will address topics including tooth brushing, denture care, inter-dental care, tongue care, and dry mouth care. There will be four sessions in total, with each intervention session lasting approximately 45 minutes.
  Arms: Interventional
Behavioral: Control Intervention — Participants will receive a home-based, un-tailored oral care training. The training includes a tooth brushing and dental care demonstration, and information about oral diseases and dry mouth. This training will be 15 minutes in duration. Participants will have the opportunity to participate in the functionally tailored intervention following the end of this study.
  Arms: Control

SUMMARY:
The specific aims of this study are:

Aim 1. Develop a staged and modifiable dyadic oral care intervention to provide functionally-tailored oral care rehabilitation for community-dwelling persons with dementia (PWD) and need-based skills training their family caregivers (CGs). Based on the literature review and MCWB, a 4-week intervention with 8 modules, including universal modules (e.g., environmental changes), CG modules (e.g., cuing strategies) and modules for both PWD and CGs (e.g., oral care techniques), will be developed addressing the relevant SCT constructs (e.g., functional deficits of PWD and caregiving needs of CGs). Guided by a validated, widely-used theory of rehabilitation medicine, modules will be used alone or in combination to provide personalized, hand-on, functionally-tailored oral care rehabilitation for PWD along with skills training for CGs to match their caregiving needs. The training focus shifts from the PWD to the CG, as the independence of the PWD decreases. Semi-structured interviews with family CGs will then be conducted (until data saturation is reached) to understand their oral care needs, desired intervention approaches, and the perceived feasibility and utility of the intervention. The intervention will be revised and then pilot tested with 4 dyads, one per each of the four functional levels of the DAT.

Aim 2. Evaluate the feasibility and efficacy of the intervention in home settings through a randomized, controlled trial with 40 pairs of PWD and their primary CGs, including immediate post-intervention and 3-month follow-up. Dyads will be stratified into 4 functional levels based on the PWD's DAT score and then randomly assigned to the intervention or control (non-tailored usual care) group.

DETAILED DESCRIPTION:
This study aims to develop and evaluate a functionally-tailored oral hygiene intervention to improve oral health for community-dwelling persons with dementia, while also reducing caregiver burden and improving the care partner relationship. The study consists of two phases. First, we will develop a modularized, functionally-tailorable oral care intervention based on caregiver qualitative interviews and existing literature. The second phase will then examine the efficacy and feasibility of the intervention through a randomized controlled trial (3 intervention: 1control ratio)with 40 Persons with Dementia/caregiver dyads. Control participants will receive the standard oral hygiene education currently provided to persons with Dementia during dental care. The Intervention group will receive 4-week, dyadic, hands-on, functionally-tailored oral care intervention. We will collect data at baseline, 4-weeks, and 3 months post intervention. After data collection, the differences in the control and intervention groups in regard to their oral hygiene, behavioral symptoms during oral care, caregiver outcomes (burden, self-efficacy) and care partner relationship will be explored.

The specific aims of this study are:

Aim 1. Develop a staged and modifiable dyadic oral care intervention to provide functionally-tailored oral care rehabilitation for community-dwelling persons with dementia (PWD) and need-based skills training their family caregivers (CGs). Based on the literature review and MCWB, a 4-week intervention with 8 modules, including universal modules (e.g., environmental changes), CG modules (e.g., cuing strategies) and modules for both PWD and CGs (e.g., oral care techniques), will be developed addressing the relevant SCT constructs (e.g., functional deficits of PWD and caregiving needs of CGs). Guided by a validated, widely-used theory of rehabilitation medicine, modules will be used alone or in combination to provide personalized, hand-on, functionally-tailored oral care rehabilitation for PWD along with skills training for CGs to match their caregiving needs. The training focus shifts from the PWD to the CG, as the independence of the PWD decreases. Semi-structured interviews with family CGs will then be conducted (until data saturation is reached) to understand their oral care needs, desired intervention approaches, and the perceived feasibility and utility of the intervention. The intervention will be revised and then pilot tested with 4 dyads, one per each of the four functional levels of the DAT.

Aim 2. Evaluate the feasibility and efficacy of the intervention in home settings through a randomized, controlled trial with 40 pairs of PWD and their primary CGs, including immediate post-intervention and 3-month follow-up. Dyads will be stratified into 4 functional levels based on the PWD's DAT score and then randomly assigned to the intervention or control (non-tailored usual care) group.

Sub-Aim 2.1 Evaluate the feasibility of the intervention across four domains: acceptability, demand, implementation, and practicality. We will interview the dyads and review their daily oral care logs at both post-intervention and 3-month follow-up, assessing satisfaction with, acceptability of, and actual use of the intervention. Oral care trainers will complete intervention logs following each training session to document the extent of content delivery, diversion from the protocol, resources used, and perceptions about intervention success. Exit interviews with PWD (when possible), CGs, and trainers will be conducted to identify potential barriers, facilitators, and needed changes.

Sub-Aim 2.2 Examine the efficacy of the intervention. We hypothesize that both PWD oral hygiene and CG self-efficacy in providing oral care will show clinically significant improvements for the intervention group compared to the control group. Secondary outcomes for PWD (e.g., behavior symptoms during oral care), CGs (e.g., oral care related burden) and the dyadic relationship (e.g., the Dyadic Relationship Scale) will also be explored.

ELIGIBILITY:
Inclusion Criteria for Caregivers:

* 18 years or older
* English-speaking
* Willing to participate in the study

Exclusion Criteria for Caregivers:

* Cognitively impaired
* Blind, deaf, or severely disabled

Inclusion Criteria for Persons with Dementia

* Diagnosis of Dementia
* Age 50 years or older or 18 years or older with Huntington's Disease
* Community-dwelling
* English speaking
* Have natural teeth
* Not blind, deaf, or severely disabled
* Have a caregiver that is age equal or 18+ years old, English speaking, cognitively intact, and willing to participate in the study

Exclusion Criteria for Persons with Dementia:

* Joint replacement with a history of prosthetic joint infection
* Requires immediate dental referrals
* Have oral cancer or active oral infection or 3) is actively dying.
* Actively dying

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xi Chen, DDS, PhD, Principal Investigator — Associate Professor
Locations (1):
- UIowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Interventional
Started (7 dyads = 14 individuals in the control group, 19 dyads = 38 individuals in the study group, Total: 26 dyads = 52 individuals started at the baseline) | 7 (This is the numbers of PWD/CG dyads included in the control group at the baseline.) | 19 (This is the numbers of PWD/CG included in the study group at the baseline)
Completed (5 dyads = 10 individuals in the control group, 13 dyads = 26 individuals in the study group, Total: 18 dyads = 36 individuals completed the study) | 5 (This is the numbers of PWD/CG dyads who completed the 3-month follow-up in the control group) | 13 (This is the numbers of PWD/CG dyads who completed the 3-month follow-up in the study group)
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 0 | 2
Not completed — Unsafe home environment for research staff | 0 | 1

BASELINE CHARACTERISTICS:
Population: 26 pairs of participants with dementia (PWD) and their family caregivers (FCG) (Total=52 participants) were enrolled into the study at the baseline. A descriptive analysis was completed for PWD and FCG, respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Interventional | Total
Number analyzed (Participants) | 14 | 38 | 52
Age, Continuous [Mean (Standard Deviation); unit: year] — Population: The overall numbers of baseline participants include 7 PWD and 7 FCG (total=14) in the control group and 19 PWD and 19 FCG (total=38). However, we analyzed PWD and FCG separately. So each row included 7 participant (7 for PWD and 7 for FCG).
  year
    Participants with dementia: number analyzed (Participants) | 7 | 19 | 26
    Participants with dementia | 70.7 (15.1) | 69.7 (17.8) | 69.9 (16.8)
    Family caregiver: number analyzed (Participants) | 7 | 19 | 26
    Family caregiver | 68.0 (21.2) | 68.0 (10.3) | 68.0 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 26 PWD/CG dyads (total=52 individuals) were included in the analysis. We reported PWD's and CG's characteristics separately.
  Participants
    Participants with dementia: number analyzed (Participants) | 7 | 19 | 26
    Participants with dementia: Female | 4 | 12 | 16
    Participants with dementia: Male | 3 | 7 | 10
    Family caregivers: number analyzed (Participants) | 7 | 19 | 26
    Family caregivers: Female | 4 | 12 | 16
    Family caregivers: Male | 3 | 7 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 26 PWD/CG dyads (total=52 individuals) were included in the analysis. We reported their characteristics separately.
  Participants
    PWD: number analyzed (Participants) | 7 | 19 | 26
    PWD: American Indian or Alaska Native | 0 | 0 | 0
    PWD: Asian | 0 | 0 | 0
    PWD: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    PWD: Black or African American | 0 | 2 | 2
    PWD: White | 7 | 16 | 23
    PWD: More than one race | 0 | 0 | 0
    PWD: Unknown or Not Reported | 0 | 1 | 1
    FCG: number analyzed (Participants) | 7 | 19 | 26
    FCG: American Indian or Alaska Native | 0 | 0 | 0
    FCG: Asian | 0 | 0 | 0
    FCG: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    FCG: Black or African American | 0 | 1 | 1
    FCG: White | 7 | 17 | 24
    FCG: More than one race | 0 | 0 | 0
    FCG: Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 38 | 52

OUTCOME MEASURES:

1. Primary Outcome: Person With Dementia: Oral Hygiene
Description: We used the Debris Index (DI) of the Oral Hygiene Index (a scale of 0 to 3, with lower values indicating no debris present and higher values indicating more soft debris on the tooth. Also called plaque score) to assess PWD's oral hygiene status. We used the percentage change in plaque scores between baseline and 3 months to evaluate the effectiveness of the proposed intervention on improving PWD's oral hygiene.
Time Frame: Baseline and 3 Months
Population: The percentage change in plaque scores between baseline and 3 months was compared between the PWD in the control group and PWD in the study group. 26 PWD (7 in the control and 19 in the study group) with completed data at the baseline. A total of 18 PWD (control group=5 and study group=13) completed the study with data on this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage change in plaque scores
Groups:
- Control - PWD: Control Intervention: Participants will receive a home-based, un-tailored oral care training. The training includes a tooth brushing and dental care demonstration, and information about oral diseases and dry mouth. This training will be 15 minutes in duration. Participants will have the opportunity to participate in the functionally tailored intervention following the end of this study.
- Interventional - PWD: Study Group Intervention: Participants receive a 4-week, hands-on, functionally-tailored intervention. The intervention will address topics including tooth brushing, denture care, inter-dental care, tongue care, and dry mouth care. There will be four sessions in total, with each intervention session lasting approximately 45 minutes.
Arm/Group | Control - PWD | Interventional - PWD
Number analyzed (Participants) | 7 | 19
percentage change in plaque scores | 29.6 (32.9) | 37.3 (23.4)

2. Primary Outcome: Self-perceived Oral Care-giving Efficacy
Description: Self-perceived Oral Care-giving Efficacy scale included 19 items to assess self-perceived efficacy in providing oral care to care recipients. We assessed CG's self-perceived oral care-giving efficacy at the baseline and 3-month follow-up visit. We used the percentage change in Self-perceived Oral Care-giving Efficacy scores between the baseline and 3-month follow-up to examine the effectiveness of the proposed intervention on improving CG's oral care-giving skills. Higher scores indicate a better improvement in self-perceived efficacy.
Time Frame: Baseline and 3 Months
Population: The percentage change in Self-perceived Oral Care-giving Efficacy scores between baseline and 3 months was compared between the control and study groups. 26 FCG with complete data were included in the baseline analysis. A total of 18 completed the study with data on this outcome measure
Measure: Mean (Standard Deviation); unit: percentage change in Self-perceived Oral
Groups:
- Control - FCG: Control Intervention: Participants will receive a home-based, un-tailored oral care training. The training includes a tooth brushing and dental care demonstration, and information about oral diseases and dry mouth. This training will be 15 minutes in duration. Participants will have the opportunity to participate in the functionally tailored intervention following the end of this study.
- Interventional - FCG: Study Group: Participants receive a 4-week, hands-on, functionally-tailored intervention. The intervention will address topics including tooth brushing, denture care, inter-dental care, tongue care, and dry mouth care. There will be four sessions in total, with each intervention session lasting approximately 45 minutes.
Arm/Group | Control - FCG | Interventional - FCG
Number analyzed (Participants) | 7 | 19
percentage change in Self-perceived Oral | 12.6 (8.3) | 17.5 (24.8)

3. Secondary Outcome: Dyadic Relationship
Description: Dyadic Relationship Scale (DRS) to measure strain between the caregiver and recipient within the past month on a scale of 1 to 4. The original DRS 11 items will be used for caregivers and 10 items will be used for care recipients. High scores indicate high levels of strain and positive interaction. We used the percentage change in dyadic relationship scores between the baseline and 3 months to examine how this intervention affected PWD/CG relationships.
Time Frame: Baseline and 3 Months
Population: The percentage change in dyadic relationship scores between baseline and 3 months was compared between the control and study groups. 12 dyads with missing data at the baseline were eliminated from the analysis. A total of 8 dyads completed the study with data on this outcome measure
Measure: Mean (Standard Deviation); unit: percentage change in dyadic relationship
Groups:
- Control - PWD/FCG Dyad: Control Group: Participants will receive a home-based, un-tailored oral care training. The training includes a tooth brushing and dental care demonstration, and information about oral diseases and dry mouth. This training will be 15 minutes in duration. Participants will have the opportunity to participate in the functionally tailored intervention following the end of this study.
- Interventional - PWD/FCG Dyad: Study Group: Participants receive a 4-week, hands-on, functionally-tailored intervention. The intervention will address topics including tooth brushing, denture care, inter-dental care, tongue care, and dry mouth care. There will be four sessions in total, with each intervention session lasting approximately 45 minutes.
Arm/Group | Control - PWD/FCG Dyad | Interventional - PWD/FCG Dyad
Number analyzed (Participants) | 4 | 11
percentage change in dyadic relationship | -10.7 (20.3) | 14.1 (27.1)

ADVERSE EVENTS:
Time Frame: 3 months
Description: The Adverse Events data were collected for PWD only.
Arm/Group | Control | Interventional
All-Cause Mortality (participants affected / at risk) | 0/5 | 2/13
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/13
Other Adverse Events (participants affected / at risk) | 0/5 | 0/13

LIMITATIONS AND CAVEATS:
We are not able to reach the targeted recruitment goal because of the impact of COVID. Therefore, this trial was inadequately powered to detect the potential differences between the study group and the control group in all of the outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT04238520/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT04238520/SAP_001.pdf
  • Informed Consent Form (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT04238520/ICF_002.pdf